CLINICAL TRIAL: NCT01460407
Title: Effect of Clarithromycin on the Pharmacokinetics of LY2216684 in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Clarithromycin on LY2216684
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14401; H9P-EW-LNEB (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-03

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2216684 + Clarithromycin (Experimental): Participants will receive a single 18-mg oral dose of LY2216684 on Days 1 and 10. Clarithromycin (500 mg) will be administered twice a day (BID) on Days 6 through 13.
  Interventions: Drug: LY2216684; Drug: Clarithromycin

INTERVENTIONS:
Drug: LY2216684 — Administered orally
Drug: Clarithromycin — Administered orally

SUMMARY:
The study will evaluate the effect of Clarithromycin on the pharmacokinetics (PK) of LY2216684 in healthy participants. Side effects will be documented. There will be 2 study periods (5 and 9 days) and follow up will occur at least 7 days after the last dose. Screening is required within 45 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical history and physical examination
* Male participants:

  o Agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug
* Female participants:

  o Are women of child-bearing potential who test negative for pregnancy at the time of enrollment, have used a reliable method of birth control (not including hormonal contraceptives) for 4 weeks prior to administration of study drug, and agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug; or women not of child-bearing potential due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation/occlusion) or menopause [at least 1 year without menses or 6 months without menses and a follicle stimulating hormone (FSH) >40 milli-international units per milliliter (mIU/mL)]
* Have a body weight >50 kilograms (kg)
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow for blood sampling as per the protocol
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the institutional review board (IRB) governing the site
* Have normal blood pressure (BP) and pulse rate (PR) (sitting position) as determined by the investigator
* Are predicted to have both cytochrome P450 (CYP)2D6 and CYP2C19 extensive metabolizer (EM) phenotypes as determined by genotyping assessment

Exclusion Criteria:

* Are currently enrolled in, have completed or discontinued within the last 30 days from a clinical trial involving an investigational product or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies/intolerance to LY2216684 or clarithromycin, related compounds, or any components of the formulation
* Are persons who have previously received the investigational product in this study, have completed or withdrawn from this study or any other study investigating LY2216684 within 6 months prior to screening
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history of/or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have a history or show evidence of significant active neuropsychiatric disease or have a history of suicide attempt or ideation
* Have a documented or suspected history of glaucoma
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Are women with a positive pregnancy test or women who are lactating
* Intend to use over-the-counter or prescription medication within 14 days prior to dosing unless deemed acceptable by the investigator and Sponsor's medical monitor. Exceptions include influenza vaccinations, the use of topical medication (provided there is no evidence of chronic dosing with the risk of systemic exposure), occasional use of acetaminophen/paracetamol/ibuprofen, hormone replacement therapy including thyroid replacement (stable dose for at least 1 month)
* Use of known inhibitors and/or inducers of CY2D6, CYP2C19, and/or CYP3A 30 days prior to enrollment or are unwilling to avoid them during the study (except for use of clarithromycin)
* Have donated blood of more than 500 mL within the last month
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), or are unwilling to stop alcohol consumption 48 hours prior to dosing in Period 1 until discharge [1 unit = 12 oz (ounces) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits]
* Consume 5 or more cups of coffee (or other beverages or foods of comparable caffeine content) per day, on a habitual basis, or are unwilling to stop caffeine consumption from 48 hours prior to dosing in Period 1 until discharge
* Participants unwilling to adhere to the smoking restrictions of the Clinical Research Unit (CRU) while a resident of the CRU
* Have consumed grapefruit or grapefruit-containing products, starfruit, or pomegranates 30 days prior to enrollment or are unwilling to avoid them during the study
* Participants determined to be unsuitable by the investigator for any reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2216684: LY2216684: a single 18-milligram (mg) tablet on Day 1
- LY2216684 and Clarithromycin: LY2216684: a single 18-mg tablet on Day 10
  Clarithromycin: 500-mg tablet twice daily on Day 6 through Day 13
Period: Period 1: Day 1 to Day 5
Arm/Group | LY2216684 | LY2216684 and Clarithromycin
Started | 14 | 0
Completed | 14 | 0
Not Completed | 0 | 0
Period: Period 2: Day 6 to Day 14
Arm/Group | LY2216684 | LY2216684 and Clarithromycin
Started | 0 | 14
Completed | 0 | 13
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: LY2216684: a single 18-mg tablet on Day 1 and Day 10
  Clarithromycin: 500-mg tablet twice daily on Day 6 through Day 13
Arm/Group | Entire Study Population
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity (AUC0-∞) of LY2216684
Description: AUC0-∞ of LY2216684 was calculated during Period 1, when 18-mg LY2216684 was administered alone and Period 2, when Clarithromycin was coadministered with LY2216684. The outcome was presented as geometric Least Squares (LS) mean and the 90% Confidence Interval (CI). Geometric LS mean was controlled by participant and treatment.
Time Frame: Predose up to 96 hours post administration of LY2216684 (Day 1) and LY2216684 + Clarithromycin (Day 10)
Population: Full Analysis Set: Participants who received at least 1 dose of LY2216684.
Measure: Geometric Mean (90% Confidence Interval); unit: nanogram*hours per milliliter (ng*h/mL)
Groups:
- LY2216684: LY2216684: a single 18-mg tablet on Day 1
Arm/Group | LY2216684 | LY2216684 and Clarithromycin
Number analyzed (Participants) | 14 | 14
nanogram*hours per milliliter (ng*h/mL) | 582 [498 to 681] | 746 [638 to 873]
Statistical Analysis 1: Comparison: LY2216684 vs LY2216684 and Clarithromycin; Test type: Superiority or Other; Ratio of geometric LS mean = 1.28, 90% CI 2-sided [1.16 to 1.42] — Ratio of LY2216684 and Clarithromycin to LY2216684

2. Primary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax) of LY2216684
Description: Cmax of LY2216684 was calculated during Period 1, when 18-mg LY2216684 was administered alone, and Period 2, when Clarithromycin was coadministered with LY2216684. The outcome was presented as geometric LS mean and the 90% CI. Geometric LS mean was controlled by participant and treatment.
Time Frame: Predose up to 96 hours post administration of LY2216684 (Day 1) and LY2216684 + Clarithromycin (Day 10)
Population: Full Analysis Set: Participants who received at least 1 dose of LY2216684.
Measure: Geometric Mean (90% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Arm/Group | LY2216684 | LY2216684 and Clarithromycin
Number analyzed (Participants) | 14 | 14
nanograms per milliliter (ng/mL) | 52.58 [46.38 to 59.61] | 63.55 [56.06 to 72.04]
Statistical Analysis 1: Comparison: LY2216684 vs LY2216684 and Clarithromycin; Test type: Superiority or Other; Ratio of geometric LS mean = 1.21, 90% CI 2-sided [1.12 to 1.31] — Ratio of LY2216684 and Clarithromycin to LY2216684

3. Primary Outcome: Pharmacokinetics: Time to Maximum Plasma Concentration (Tmax) of LY2216684
Description: Tmax of LY2216684 was calculated during Period 1, when 18-mg LY2216684 was administered alone, and Period 2, when Clarithromycin was coadministered with LY2216684. The outcome was presented as geometric LS mean and the 90% CI. Geometric LS mean was controlled by participant and treatment.
Time Frame: Predose up to 96 hours post administration of LY2216684 (Day 1) and LY2216684 + Clarithromycin (Day 10)
Population: Full Analysis Set: Participants who received at least 1 dose of LY2216684.
Measure: Median (90% Confidence Interval); unit: hours (h)
Arm/Group | LY2216684 | LY2216684 and Clarithromycin
Number analyzed (Participants) | 14 | 14
hours (h) | 2.00 [1.00 to 5.00] | 2.00 [2.00 to 4.00]
Statistical Analysis 1: Comparison: LY2216684 vs LY2216684 and Clarithromycin; Test type: Superiority or Other; p = 0.7656, Wilcoxon (Mann-Whitney); Median of paired differences = 0.00, 90% CI 2-sided [-0.50 to 0.50] — LY2216684 and Clarithromycin minus (-) LY2216684

ADVERSE EVENTS:
Description: All randomized participants were to receive the following treatment regimen:
  LY2216684: a single 18-mg tablet on Day 1 and a single 18-mg tablet on Day 10
  Clarithromycin: 500-mg tablet twice daily on Day 6 through Day 13
Groups:
- LY2216684: Adverse Events (AEs) that occurred from Day 1 postdose to Day 6 prior to dosing for all randomized participants.
- LY2216684 and Clarithromycin: AEs that occurred from Day 10 postdose to end of study (7 days post last dose) for all randomized participants.
- Clarithromycin: AEs that occurred from Day 6 postdose to Day 10 prior to dosing, for all randomized participants.
Arm/Group | LY2216684 | LY2216684 and Clarithromycin | Clarithromycin
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 6/14 | 6/14 | 4/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2216684 (N=14) | LY2216684 and Clarithromycin (N=14) | Clarithromycin (N=14)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Penile discharge (Reproductive system and breast disorders) | 0/8 (0) | 2/8 (2) | 0/8 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days